CLINICAL TRIAL: NCT03678415
Title: Community Based Maternal Healthcare Services
Brief Title: Package of Community-based Mental Healthcare Services in Preventing Perinatal Mental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR-17042
Record Dates: First submitted 2018-06-11; First posted 2018-09-19 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2018-06

CONDITIONS: Mental Disorder
Keywords: Depression, anxiety and stress
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders | interventions — Drug Packaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control (Experimental): In the control arm, the community healthcare providers serve usual health education like counseling as they provided in perinatal period of enrolled mothers regular follow up basis. This health education is different from developed intervention. But service provider does not know. The investigators select community clinic before provide training regarding training manual. For this, the investigators selected 11 cluster randomly among the 23 community clinics' in the primary health care in study area and provide common health education instructions to the enrolled mothers. But service providers does not know the intervention package services that will provide in intervention arm's service providers.
  Interventions: Behavioral: Community-Based Primary Mental Health Care (CBPMHC) package

INTERVENTIONS:
Behavioral: Community-Based Primary Mental Health Care (CBPMHC) package — According to the intervention package, after receiving training, the service providers will start providing service according to learning to the enrolled mothers. The intervention package has developed in many maternal and psychosocial supports like psycho-educational communication about pregnancy complications, danger signs, birth preparedness; psycho-social support including information about psycho-education, graded activities and different types of alternative thoughts. Besides, in this regard the investigators included anxiety and depression disorders symptoms, postpartum mood disorders like postpartum blue, postpartum psychosis, etc. The primary healthcare service provider's provide intervention along with their daily routine and investigators follow it up by their visits.

SUMMARY:
During pregnancy and in the year after birth women can be affected by a range of mental health problems. Anxiety and depression are the most prevalent mental illnesses during the perinatal period. In low socio-economic country like Bangladesh, there is a huge knowledge gap. Perinatal mental disorders are preventable or manageable conditions if can be addresses primariliry at the community level. Better antenatal detection of depression offers an opportunity for earlier intervention to address the illness and reduce the risk that will cause longer term problems for the mother or her baby. Most of the patients do not seek care for mental health problems as they think if they go for treatment other people would tell them 'mad'. Moreover, due to lack of necessary training of the healthcare providers at primary and secondary level the patients with mental health problems cannot get adequate services to meet the requirements. Objective of the study is to develop a package of community-based primary mental healthcare services for delivering with the maternal services care in preventing perinatal mental disorders.

The investigators will conduct an interventional study by using both quantitative and qualitative research methodology. At first, a literally feasible package of community-based primary mental healthcare services will be developed through series of workshops. Then training will be provided to the community health workers on developed package. For the cluster randomization trial will be done to test the efficacy in reduction of perinatal mental disorders. One group of pregnant mothers will be provided the developed package of sevices along with the antenatal care and another group will be provided only routine antenatl care. Both the groups will be ensured at least four sessions of antenatal care. Following up will be through the whole pregnancy period. Afterthat, assessment will be done on mental disorders (anxiety and depression) among the both groups and will be compared to find the efficacy of the package in terms of proportion of mental disorders among the perinatal mothers. For data collection, we use different check list. Moreover, in-depth interview and focus group discussion with different groups of community people will be done to get feedback and suggestions on the package. Then the community based primary mental healthcare package will be finalized.

DETAILED DESCRIPTION:
Globally mental health conditions are of rising concern due to increased contribution to the global burden of disease. Mental health wellbeing cannot be determined by only the absence of mental disorders but also determined by related socio-economic, biological and environmental factors. Mental health disorders refer to a set of medical conditions that affect a person's thinking, feeling, mood, ability to relate to others, and daily functioning. According to the World Health Organization mental disorders comprise a broad range of problems, with different symptoms.

Depression is the most prevalent mental illness in the perinatal period, with research suggesting that around 10 to 14% of mothers are affected during pregnancy or after the birth of a baby. The key symptoms of depression include persistent sadness, fatigue and a loss of interest and enjoyment in activities. A number of studies have shown that many women who have postnatal depression have symptoms of depression in pregnancy, and can be identified in antenatal period. Better antenatal detection of depression therefore offers an opportunity for earlier intervention to address the illness and reduce the risk that will cause longer term problems for the mother or her baby.

Public services are failing to tackle perinatal mental disorders effectively due to lack of mental healthcare providers. To achieve Sustainable Development Goal (SDG), mental health services must be available at the community level in low socioeconomic country like Bangladesh. Moreover, due to lack of necessary training the healthcare providers at primary and secondary level, the patients with mental health problems cannot get adequate services to meet the requirements. Again they fail to refer the severely ill patients to the appropriate referral centre. Mental health issues are the vital for maintaining quality of life of people in developing countries like Bangladesh.

In Bangladesh there is a strong community-based healthcare network such as union health and family welfare centers at the union levels, community clinics at community levels to provide essential healthcare services especially for mother and child. Along with this the community health workers also provide maternal services through satellite clinics, out-reach centers and home visit. It is evidenced that community based intervention like counseling and psycho-social therapy by the non-mental health specialists such as community health workers compared to the usual maternal care is associated with the reduction of symptoms of common perinatal mental disorders. So, maternal healthcare services are the appropriate ones for providing primary mental healthcare services. There is needed to provide basic mental healthcare services along with maternal healthcare services from the community level health centers as well as by the community health workers for improving perinatal mental health status in Bangladesh. Objectives of this study are a) to develop a draft package of community-based primary mental healthcare services, b) to find the feasibility of the developed package for delivering with the maternal care services, c) to test the efficacy of the package of community-based primary mental healthcare services and d) to document the healthcare seeking behavior for perinatal mental disorders.

Methods The investigators will conduct a mixed method study to develop a package of community-based primary mental healthcare services (CBPMHC). Initially a draft package of services will be developed. Then, piloting will be done as cluster randomized control trial to test the efficacy of the package. The draft CBPMHC services package will be the intervention.

The study will take place at Sadar Upazila (sub district) of Rajbari district in Bangladesh. The upazila consists of 14 unions and 294,701 populations. There are one upazila health complex, 34 community clinics, 42 health assistants and 45 family welfare assistants in the upazila. Moreover, for the qualitative part of the study additional two groups i.e community healthcare provider and community stakeholders will be the study population.

i) Development of draft package of community-based primary mental healthcare services as intervention The investigators will conduct multi-stakeholder consultative workshops at national and local level by engaging the professional bodies (psychologists, psychiatrists, and obstetricians), health program mangers, researchers and policy makers, community health workers; community stakeholders etc. A training module will also be developed related to this package.

Description of the package The package will consist of psycho-educational communication about pregnancy complications, danger signs, birth preparedness; psycho-social counseling including information about the risk factors for developing perinatal mental disorders; a psychological component and strategies (e.g. increasing positive thinking and pleasant activities, improving self-esteem and self-care) etc.

ii) Cluster randomized trial Cluster randomized controlled trial will be done to test the efficacy of the CBPMHC package. The unit of assignment will be the cluster which will be defined as the catchment areas of each community clinic. Among all the clusters in the study upazila, 22 clusters will be selected randomly for control trial. Again randomization will be done among the selected 22 clusters to assign each 11 clusters in intervention group and control group. Then required number of pregnant mothers will be enrolled as intervention group and control group. The trained community health workers will deliver the package of community mental healthcare services to the pregnant women of intervention group along with the routine maternal care.

Sampling The investigators used incidence of depression among 23.4% mother in rural Bangladesh found in a population based study. It was assumed that it will be decreased up to 15.7% that means difference between intervention and control group will be about 7.7 and intra-cluster correlation of 0.006. Sampling was estimated according to the calculation of fixed numbered clusters with flexible cluster size. Thus for a two-arm cluster randomized trial, where a minimum number of cluster is 11 in each arm, minimum 55 respondents per cluster is required at 80% power and 95% CI and 5% precession by using the following formula n= {2(Zα/2 + Zβ) 2 P (1-P)}/( P1 - P2) 2 Where, n = sample size, P1=incidence of outcome in comparison group= 0.234 P2= incidence of outcome in intervention group= 0.157 P= Pooled incidence = (P1+ P2)/2 Zα/2 = 1.96 (for α= 0.05 for 95% confidence interval) Zβ = 0.84 (for β = 0.20 for 80% power) So, the number of sample is (55x11)=605 participants in each arm and total number of sample size is 1210.

Inclusion criteria of the study participants

* Permanent resident of the study area
* Pregnant women aged >18 years
* Upon taking informed consent Exclusion criteria from the study
* Temporary resident of the study areas
* Severely ill patients (documented by registered physician with prescription)
* Refusal to take part in the study Intervention Pregnant women of first trimester will be enrolled as study participants through home visit. The trained community health workers will provide CBPMHC package of services to the mothers of the intervention arm during each routine antenatal care (at least 4) ANC visit. The pregnant women of the control arm will be provided only routine antenatal care. The intervention period will be whole pregnancy period.

Data collection: Socio-demographic and obstetric characteristics will be collected from all the study participants using semi-structured questionnaire. Mental health status (anxiety and depression) of the participants will be measured by using Bangle validated tools such as Edinburgh Postnatal Depression Scale (EPDS) rating scale is (0) for as much as I always could, (1) for not quite so much now, (2) for definitely not so much now, (3) for not at all, for depression, postnatal blue and Depression, Anxiety and Stress Scale (DASS), and rating scale is (0) for did not apply to me at all, (1) for applied to me to some degree, or some of the time, (2) for applied to me to a considerable degree, or a good part of time, (3) for applied to me very much, or most of the time for anxiety. Then another assessment on mental health status will be done among the both groups of mothers. icddr,b field team will collect data through visiting the mothers at their households. Comparison will be done between the intervention and control groups to find the efficacy of the developed package of primary mental healthcare services.

Follow-up and monitoring: During the implementation of the study periodic monitoring and supporting supervision will be continuing. The service delivery will be supervised and monitored by an efficient team. Follow-up of the pregnant women will be done along with motivation for getting at least 4 antenatal care visits. Community support groups existed surrounding the community clinics will be engaged in motivating the pregnant women coming at the community clinics for antenatal care visits. Also check-list will be used for keeping record.

Data Analysis: All the data of both intervention and control groups will be entered in the computer and necessary cleaning, editing and collation will be done. Data will be analyzed by using SPSS software (Version 21.0). Descriptive statistics will include frequency, mean, median and SD. To find out efficacy of the intervention relevant test of significance (both parametric and non-parametric) will be done. Socio-demographic characteristics will consider. Association between socio-demographic characteristics and the perinatal disorders will be tested by using chi-square test and logistic regression by considering total score as for DASS, (0-7) is normal, (8-9) is mild, (10-14) is Moderate, (15-19) is severe and 20+ is extreme to measuring anxiety. And EPDS for depression while less than 8 for depression not likely, 9-11 for depression possible, 12-13 for Fairly high possibility of depression and 14 and higher for probable depression iii) Qualitative data collection and analysis: For documentation of healthcare seeking behavior for perinatal mental disorders, the investigators obtain data by using in-depth interview (IDI) and focus group discussion (FGD). All the tape recorded interviews and interview-notes will then be placed in organized transcripts. After reviewed transcription, the investigators will use Atlas ti 5.2 software for analysis. Triangulation and analyses will be done manually.

iv) Limitation of the study: As there is time constraint and limitation of fund the follow-up period has been shortened. But this study will generate knowledge on the effect of community based mental healthcare package for reduction of anxiety and depression symptoms among the mothers.

v) Ethical Assurance for Protection of Human rights Ethical clearance has been obtained from the institutional review board (IRB) of icddr,b. The Ethical review committee follows international ethical standards to ensure confidentiality, anonymity, and informed consent. Enrollment in the study will be done only after obtaining informed consent. The investigator will assure to the participant's information use will safe form bad uses.

ELIGIBILITY:
Inclusion Criteria:

* Permanent resident of the study area
* Pregnant women aged >18 years
* Upon taking informed consent

Exclusion Criteria:

* Temporary resident of the study areas
* Severely ill patients (documented by registered physician with prescription)
* Refusal to take part in the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1210 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Number of study participants with depression, anxiety and stress in perinatal period | 18 months
  Investigators assume developed intervention helps to prevent mental health disorders

SECONDARY OUTCOMES:
Number of live births among the study participant's fetus | 18 months
  Developed intervention helps to increase live births among the study participant's fetus
Number of still births among the study participant's fetus | 18 months
  Developed intervention helps to decrease still births among the study participant's fetus
Number of low birth weight babies among the study participant's fetus | 18 months
  Developed intervention helps to decrease still births among the study participant's fetus

CONTACTS AND LOCATIONS:
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Result] Gruebner O, Khan MM, Lautenbach S, Muller D, Kramer A, Lakes T, Hostert P. Mental health in the slums of Dhaka - a geoepidemiological study. BMC Public Health. 2012 Mar 9;12:177. doi: 10.1186/1471-2458-12-177. PMID 22404959
- [Result] Hossain MD, Ahmed HU, Chowdhury WA, Niessen LW, Alam DS. Mental disorders in Bangladesh: a systematic review. BMC Psychiatry. 2014 Jul 30;14:216. doi: 10.1186/s12888-014-0216-9. PMID 25073970
- [Result] Deuchar N. New Joint Commissioning panel for mental health could help GPs to commission mental health services more effectively. Ment Health Today. 2011 Jun:9. No abstract available. PMID 21850743
- [Result] Oates M. Perinatal maternal mental health services. Recommendations for provision of services for childbearing women. London: Royal College of Psychiatrists. 2001
- [Result] O'Hara MW, Swain AM. Rates and risk of postpartum depression - a meta-analysis. Int Rev Psychiatry, 1996; 8:37-54
- [Result] Teixeira C, Figueiredo B, Conde A, Pacheco A, Costa R. Anxiety and depression during pregnancy in women and men. J Affect Disord. 2009 Dec;119(1-3):142-8. doi: 10.1016/j.jad.2009.03.005. Epub 2009 Apr 5. PMID 19346001
- [Result] Heron J, O'Connor TG, Evans J, Golding J, Glover V; ALSPAC Study Team. The course of anxiety and depression through pregnancy and the postpartum in a community sample. J Affect Disord. 2004 May;80(1):65-73. doi: 10.1016/j.jad.2003.08.004. PMID 15094259
- [Result] Josefsson A, Berg G, Nordin C, Sydsjo G. Prevalence of depressive symptoms in late pregnancy and postpartum. Acta Obstet Gynecol Scand. 2001 Mar;80(3):251-5. doi: 10.1034/j.1600-0412.2001.080003251.x. PMID 11207491
- [Result] Ramchandani P, Stein A, Evans J, O'Connor TG; ALSPAC study team. Paternal depression in the postnatal period and child development: a prospective population study. Lancet. 2005 Jun 25-Jul 1;365(9478):2201-5. doi: 10.1016/S0140-6736(05)66778-5. PMID 15978928
- [Result] Ramchandani PG, Psychogiou L, Vlachos H, Iles J, Sethna V, Netsi E, Lodder A. Paternal depression: an examination of its links with father, child and family functioning in the postnatal period. Depress Anxiety. 2011 Jun;28(6):471-7. doi: 10.1002/da.20814. Epub 2011 Apr 19. PMID 21506206
- [Result] Edge D. Perinatal Mental Health of Black and Minority Ethnic Women: A Review of Current Provision in England, Scotland and Wales. National Mental Health Development Unit. 2011.
- [Result] Center on the Developing Child at Harvard University. Maternal Depression Can Undermine the Development of Young Children: 2009; Working Paper No. 8
- [Result] World Health organization. Health in 2015: from MDGs, Millennium Development Goals to SDGs, Sustainable Development Goals. WHO 2015
- [Result] Clarke K, King M, Prost A. Psychosocial interventions for perinatal common mental disorders delivered by providers who are not mental health specialists in low- and middle-income countries: a systematic review and meta-analysis. PLoS Med. 2013 Oct;10(10):e1001541. doi: 10.1371/journal.pmed.1001541. Epub 2013 Oct 29. PMID 24204215
- [Result] Nasreen HE, Edhborg M, Petzold M, Forsell Y, Kabir ZN (2015) Incidence and Risk Factor of Postpartum Depressive Symptoms in Women: A Population Based Prospective Cohort Study in a Rural District in Bangladesh. J Depress Anxiety 4 (2): 1000180
- [Result] Morrell CJ, Warner R, Slade P, Dixon S, Walters S, Paley G, Brugha T. Psychological interventions for postnatal depression: cluster randomised trial and economic evaluation. The PoNDER trial. Health Technol Assess. 2009 Jun;13(30):iii-iv, xi-xiii, 1-153. doi: 10.3310/hta13300. PMID 19555590
- [Derived] Dutta GK, Ahmed HU, Talukder MQ, Bhattacharyya DS, Reza MS, Rahman MM, Majumdar R, Tofail F, Perry HB, Biswas TK. Effectiveness of a package of community-based mental healthcare services to address perinatal mental disorders in Bangladesh: A cluster-randomized controlled trial. Asian J Psychiatr. 2024 Dec;102:104290. doi: 10.1016/j.ajp.2024.104290. Epub 2024 Oct 25. PMID 39500096